CLINICAL TRIAL: NCT02836834
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of Recombinant Humanized Anti-PD-1 Monoclonal Antibody for Injection in Patients With Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics & Pharmacodynamics of an Anti-PD-1 mAb for Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-YKZL-I
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Lymphoma; Lung Cancer
Keywords: immunotherapy; check point inhibitor; PD-1 antibody; solid tumor; lymphoma; phase 1 trial
MeSH Terms: conditions — Lymphoma; Lung Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Escalation Cohort (Experimental): JS001
  Interventions: Biological: JS001
- Expanded cohort 1 (Experimental): The subjects of expanded cohort 1 will use repeated doses every 2 weeks like multiple dose cohorts
  Interventions: Biological: JS001
- Expanded cohort 2 (Experimental): The subjects of expanded cohort 2 will use repeated doses every 2 weeks like multiple dose cohorts
  Interventions: Biological: JS001

INTERVENTIONS:
Biological: JS001 — Dose escalation study evaluating three dose levels (1, 3 and 10 mg/kg) of JS-001.Each of the 3 dose levels will use 2 dose schedules: single dose, and repeated doses every 2 weeks. Subjects will be assigned to a dose schedule in the order of study entry.
  Other Names: toripalimab, TAB001

SUMMARY:
The primary objective is to assess the safety and tolerability of JS-001 in subjects with various advanced or recurrent malignancies, including solid tumors and lymphomas, and to evaluate its preliminary efficacy.

The secondary objectives are to: 1) characterize the single-dose and multi-dose pharmacokinetic (PK) profile of JS-001, 2) characterize the immunogenicity of JS-001; 3) assess the dose-efficacy relationship of JS-001 single agent, and 4) preliminarily evaluate biomarkers associated with the efficacy of JS-001.

The exploratory objectives include to evaluate the consistency between biomarker detection results of archived tissue and fresh frozen tissue, and to assess the consistency of response using various response criteria (such as irRC, WHO, RECIST and irRECIST).

DETAILED DESCRIPTION:
OVERVIEW This is a Phase 1, open-label, dose-escalation study of JS-001, a humanized monoclonal IgG4 antibody targeting the Programmed Death -1 (PD-1). It is estimated that 18-36 subjects with advanced or recurrent solid tumors or lymphomas will be enrolled in the dose-escalation study.

A 3+3 design will be utilized for this Phase 1 study. Three dose levels are planned and include: 1, 3, 10 mg/kg/dose. Each of the 3 dose levels will use 2 dose schedules: single dose, and repeated doses every 2 weeks. Subjects will be assigned to a dose schedule in the order of study entry.

The study will be the traditional 3 + 3 design with 3 or 6 subjects treated at this dose level and at all subsequent dose levels depending upon the incidence of DLTs. If no DLTs occur in a cohort of 3 subjects, a new cohort of 3 subjects will be treated at the next higher dose level. If 1 of 3 subjects in a cohort experiences a DLT, that cohort will be expanded to 6 subjects. If only 1 of the 6 subjects has a DLT, then the next cohort of 3 subjects will be treated at the next higher dose level. If 2 or more DLTs occur within a cohort, then that dose level will be above the MTD (the highest dose where no more than 1 of 6 subjects has experienced a DLT), and the previous lower (tolerated) dose level will be considered the MTD.

A DLT is defined as a Grade 3 drug-related adverse event occurring within 28 days after previous dose (excluding tumor flare defined as local pain, irritation, or rash localized at sites of known or suspected tumor or a transient Grade 3 infusion adverse event) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 in a single dose cohort.

Tumor response will be evaluated using immune-related response criteria (irRC), , Response Evaluation Criteria in Solid Tumors (RECIST 1.1), , and International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphomas (for lymphomas only).

In the absence of confirmed disease progression and intolerable toxicities, subjects in the single dose cohorts and multiple dose cohorts will be allowed to continue JS-001 administration with the consent of the subject.

If there is an effective case in a given dose level and the safety is good (There is no more than Grade 2 adverse event (not included Grade 2), 6-14 subjects with soft tissue sarcoma will be enrolled in the dose level as expanded cohort. The subjects of expanded cohort will use repeated doses every 2 weeks like multiple dose cohorts to further evaluate safety and efficacy of JS-001 with soft tissue sarcoma. At the same time, 9-12 subjects with hodgkin lymphoma will be enrolled in 3 mg/kg/dose level as expanded cohort. The subjects of expanded cohort will use repeated doses every 2 weeks like multiple dose cohorts to further evaluate safety and efficacy of JS-001 with hodgkin lymphoma.

DOSAGE AND ADMINISTRATION JS-001 will be administered as a 60-minute i.v. infusion. Cohorts will include escalating dose levels of 1, 3, 10mg/kg/dose.

SAFETY EVALUATIONS Assessment of safety will be determined by vital sign measurements, clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status evaluations, diagnostic imaging, physical examinations, electrocardiograms, and the incidence and severity of adverse events.

Safety will also include evaluations of immune safety and immunogenicity. Particular attention will be given to adverse events that may follow enhanced T-cell activation such as dermatitis and colitis, uveitis, or other immune-related adverse events (irAEs).

An irAE is a clinically significant adverse event of any organ that is associated with drug exposure, of unknown etiology, and is consistent with an immune-mediated mechanism.

EFFICACY EVALUATIONS The primary efficacy endpoint is the best response rate (RR). Duration of response, progression-free survival, time to progression, and overall survival will also be analyzed.

PHARMACOKINETIC EVALUATIONS Pharmacokinetic parameters include AUC, Cmax, tmax, and t½, etc. STATISTICAL METHODS The sample size for this study is not determined from power analysis. It is based on the 3+3 design for dose escalation and safety evaluation requirements.

Descriptive statistics will include: mean, standard deviation, median, and minimum and maximum values for continuous variables; frequencies and percentages for categorical variables.

The efficacy parameters will be summarized using descriptive statistics. All safety and pharmacokinetic parameters will be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign Informed Consent;
2. Re-entry into the study is allowed with a second informed consent;
3. Willing to provide blood sample for biomarker analysis(mandatory). The tissue sample is optional;
4. A diagnosis of an advanced malignant tumor confirmed by histology or cytology;
5. No standard of care for the patient;
6. At least 1 measurable lesion;
7. Aged 18-65 years;
8. Anticipated life expectancy of at least 3 months;
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
10. i) At least 4 weeks elapsed since receiving systemic chemotherapy, at least 6 weeks since receiving mitomycin or nitrosoureas, and at least 2 weeks since receiving a tyrosine kinase inhibitor;
11. At least 4 weeks elapsed since receiving definite radiotherapy, and at least 2 weeks since receiving palliative radiotherapy;
12. At least 2 weeks since the last dose of systemic steroid therapy (>10 mg/day prednisone or equivalent);
13. At least 4 weeks since receiving anti-cancer biotherapy;
14. Recovered from previous treatment related adverse reaction;
15. willing to use an acceptable contraceptive method;
16. A negative pregnancy test for female subjects of childbearing potential;

Exclusion Criteria:

1. Active central nervous system (CNS) metastases and/or carcinomatous meningitis;
2. Known history of another primary solid tumor, unless the participant has undergone potentially curative therapy with no evidence of that disease for 2 years, or underwent successful definitive resection of basal or squamous cell carcinoma of the skin, or in situ cervical cancer;
3. Active, known or suspected autoimmune disease;
4. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2,or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) blocking antibodies;
5. Significant medical disease;
6. Active infection;
7. Active tuberculosis or history of tuberculosis with one year;
8. Infection of Human immunodeficiency virus (HIV);
9. A complication requiring immune-suppression;
10. Received a live vaccine within 4 weeks prior to first dose of study drug
11. pleural or abdominal effusion with symptoms;
12. Drug or alcohol abuse (for subjects in the pharmacokinetic cohorts) ;
13. evidence of interstitial lung disease;
14. Active hepatitis B or C, or with significant risk of hepatitis reactivation;
15. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to monoclonal antibodies or drugs chemically related to the study drug. History of serious hypersensitivity reaction or serious hepatotoxicity related to any drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 154 days

SECONDARY OUTCOMES:
correlation analysis of PD-L1 expression of tumor and ORR | 154 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, PhD.MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang J, Dong L, Yang S, Han X, Han Y, Jiang S, Yao J, Zhang Z, Zhang S, Liu P, Qin Y, Wu H, Feng H, Yao S, Sun Y, Song H, Shi Y. Safety and clinical efficacy of toripalimab, a PD-1 mAb, in patients with advanced or recurrent malignancies in a phase I study. Eur J Cancer. 2020 May;130:182-192. doi: 10.1016/j.ejca.2020.01.028. Epub 2020 Mar 27. PMID 32224416